CLINICAL TRIAL: NCT00216450
Title: An Open Observational Study For The Rabeprazole Administration In Adult Subjects With Helicobacter Pylori (H. Pylori) Infection
Brief Title: Study of the Safety and Effectiveness of Rabeprazole in Treatment of Helicobacter Pylori Infection in Adults.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Cilag Pharmaceutica S.A.C.I., Greece (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003478
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Helicobacter Infections; Bacterial Infections
Keywords: rabeprazole; proton pump inhibitor; Helicobacter infections; Helicobacter pylori; H pylori; bacterial infections
MeSH Terms: conditions — Helicobacter Infections; Bacterial Infections | interventions — Rabeprazole

INTERVENTIONS:
Drug: rabeprazole sodium

SUMMARY:
The purpose of the study is to confirm the safety and effectiveness of rabeprazole in the treatment of adult patients with Helicobacter pylori (H. pylori) infection in routine clinical practice.

DETAILED DESCRIPTION:
An infection of Helicobacter pylori (H. pylori) is a risk factor for many types of gastrointestinal diseases and associated with stomach inflammation, ulcer of the stomach or small intestine. The recommended treatment for the infection is a triple therapy consisted of one proton pump inhibitor, such as rabeprazole, and two antibiotics administered for 7 days. This is an open label, nonrandomized study of the safety of rabeprazole in the treatment of patients with H. pylori infection. The study consists of 2 phases: the 2-month main phase and the 4-month monitoring phase (total duration of 6 months). During the main phase, patients are treated for 7 days with three drugs (rabeprazole, clarithromycin, and amoxycillin), and the effectiveness of the treatment is assessed 4 weeks later. During the monitoring phase, patients are interviewed at monthly intervals to assess symptoms and to report any adverse events. Safety assessments include the incidence of adverse events throughout the treatment and monitoring phases, and laboratory tests (hematology, biochemistry, urinalysis) and vital signs at the start of the study and after 1 month. Assessments of effectiveness include the eradication of H. pylori infection, assessed by the urea breath test one month after treatment. The primary study hypothesis is that rabeprazole is well-tolerated long-term in the treatment of patients with H. pylori infection in routine clinical practice. Rabeprazole tablets (20 milligrams[mg]) taken orally twice daily for 7 days. Clarithromycin (500mg) and amoxycillin (1 gram) taken twice daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Helicobacter pylori (H. pylori) infection
* patients over 45 years of age must have an endoscopic examination of the digestive system
* patients must have positive result of urea breath test (UBT) for H. pylori
* patients being treated with rabeprazole in combination with clarithromycin and amoxycillin to eradicate H. pylori.

Exclusion Criteria:

* Known hypersensitivity to rabeprazole, clarithromycin, or amoxycillin
* evidence from endoscopic examination of gastrointestinal hemorrhage or stomach cancer, or had previous stomach surgery
* use of aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), antibiotics, bismuth, or proton pump inhibitors during the last 4 weeks prior to study initiation
* history of successful treatment to eradicate H.pylori infection
* females who are pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2004-10; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events throughout the study

SECONDARY OUTCOMES:
Laboratory tests (hematology, biochemistry, urinalysis) and vital signs at start of study and one month after treatment; eradication of H. pylori infection, assessed by urea breath test one month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pharmaceutica S.A.C.I. Clinical Trial, Study Director — Janssen-Cilag Pharmaceutica S.A.C.I.